CLINICAL TRIAL: NCT00738868
Title: Re-irradiation and Stereotactic Cetuximab in Patients With Recurrent Carcinoma of the Head and Neck
Brief Title: Cetuximab and Stereotactic Radiation Therapy in Treating Patients With Recurrent Head and Neck Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000589673; COL-CKNO-RERT; COL-0705; INCA-RECF0629
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-07

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage III salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Cetuximab; Radiosurgery

INTERVENTIONS:
Biological: cetuximab
Radiation: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving cetuximab together with stereotactic radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how giving cetuximab together with stereotactic radiation therapy works in treating patients with recurrent squamous cell carcinoma of the head and neck cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate local control at 12 months in patients with recurrent squamous cell carcinoma of the head and neck treated with cetuximab and stereotactic radiotherapy.

Secondary

* Determine the incidence of cutaneous toxicity.
* Assess the care and development of skin reactions.
* Determine the quality of life of patients treated with this drug.
* Determine tumor response at 2 months.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV once weekly for 5 weeks. Patients undergo stereotactic radiotherapy 3 times weekly during weeks 2 and 3.

After completion of study therapy, patients are followed at 2 months and then every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Unresectable disease
  * Recurrent disease
* No metastatic disease
* Disease in previously irradiated area must be proven by biopsy or imaging

  * At least 3 months between prior radiotherapy and diagnosis of recurrent disease
* Surgery or brachytherapy must be possible
* Measurable or evaluable disease by RECIST criteria
* No available curative therapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Not pregnant or nursing
* No psychological, familial, social, or geographical reasons that would make monitoring the patient impossible
* No other malignant disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another clinical study of an experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with nonprogressive disease at 12 months according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lartigau, MD, PhD, Study Chair — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France